CLINICAL TRIAL: NCT02696824
Title: Effectiveness of Nurse-delivered Care for Adherence/Mood in HIV in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Massachusetts General Hospital (Other); University of Cape Town (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Steven Safren, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20150399; 1R01MH103770-01A1 (NIH)
Record Dates: First submitted 2016-02-18; First posted 2016-03-02 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Immunodeficiency Virus, Human; Depressive Symptoms
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-AD (Experimental): Those assigned to the CBT-AD [cognitive behavioral therapy for adherence and depression) condition, will have up to 8 additional sessions delivered by the study clinic nurse. Additionally, those assigned to CBT-AD will have the procedures available to those assigned to ETAU.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Adherence and Depression
- ETAU (No Intervention): Participants in both conditions receive usual care plus the following procedures below.
  All participant will have the benefit of the psychosocial assessment, and the clinic nurse will provide feedback to the participant and to their clinic doctor about their depression. Additionally, all participants will undergo standard of care "second line treatment" adherence counseling in the clinic . The clinic doctor will not be restricted in terms of referral or treatment of depression for their patient with respect to antidepressant medications or other interventions available.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Adherence and Depression — This treatment involves integrating CBT for depression with CBT for adherence following our "Life-Steps" approach.
  Arms: CBT-AD

SUMMARY:
The purpose of this study is to conduct a two-arm effectiveness trial in Cape Town, South Africa of a Xhosa-adapted, nurse-delivered, cognitive behavioral therapy (CBT) treatment for depression and adherence, integrated into the HIV care setting in patients with HIV who did not achieve viral suppression from first-line treatment. The CBT treatment will be compared to enhanced usual care (Enhanced Treatment As Usual - ETAU) on study endpoints (as described in study endpoints section below).

DETAILED DESCRIPTION:
Clinical Clinical depression is one of the highest comorbidities to HIV/AIDS, with estimated rates up to 34.9 percent. Depression, in the context of HIV, leads to poor self-care behavior such as non-adherence to ART and worse retention in care, which are critical for treatment success. Based on our prior work, and given that CBT is an evidenced-based treatment for depression, this is a two-arm effectiveness randomized controlled trial of nurse-delivered cognitive behavioral therapy for depression and adherence integrated into the HIV primary care setting in S. Africa. To ensure that those who need this intervention the most will receive it, participants will be patients with HIV who did not achieve viral suppression from their first line ART, and have a unipolar depressive mood disorder.

ELIGIBILITY:
Inclusion Criteria:

* HIV-seropositive
* Current diagnosis of depression
* Did not attain viral suppression from first-line ARV per local clinic standard

Exclusion Criteria:

* Unable or unwilling to provide informed consent.
* Active untreated, major mental illness (untreated psychosis or mania) that would interfere with CBT-AD.
* Has not received CBT for depression.
* Less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2016-07-19 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
Changes in HIV medication adherence throughout intervention phase | Assessed between baseline and the 4 month assessment
  Percentage of prescribed antiviral therapy agent (medications ) taken as measured by real time wireless motoring device
Depression scores as assessed by an independent (blind assessor) after intervention. | 4 month assessment
  Hamilton Depression Rating Scale
  The Hamilton Depression Rating Scale has a total score ranging from 0-54, with higher scores indicated greater depressive symptoms.

SECONDARY OUTCOMES:
HIV viral load | 12-month assessment
  Percentage of patients with a detectable viral load at the 12 month assessment
CD4 | 12-month assessment
  Mean CD4 cell counts at the 12 month assessment
HIV medication adherence over follow-up | Aggregate across 4,8, and 12-month assessment
  Percentage of prescribed antiviral therapy agent (medications ) taken as measured by real time wireless motoring device
Depression scores as assessed by an independent (blind assessor) over follow-up | Aggregate across 4,8, and 12-month assessment
  Hamilton Depression Rating Scale
  The Hamilton Depression Rating Scale has a total score ranging from 0-54, with higher scores indicated greater depressive symptoms.

OTHER OUTCOMES:
Depression scores via self-report after intervention | 4-month assessment
  Center for Epidemiological Studies-Depression (CES-D) scale
  The CES-D has a total score ranging from 0-60, with higher scores indicated greater depressive symptoms.
Depression scores via self-report over follow up | Aggregate across 4,8, and 12-month assessment
  CES-D scale
  The CES-D has a total score ranging from 0-60, with higher scores indicated greater depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Safren, PhD, Principal Investigator — University of Miami
Locations (3):
- United States (2):
  - University of Miami, Miami, Florida
  - The General Hospital Corp dba Massachusetts General Hospital, Boston, Massachusetts
- University of Cape Town, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Safren SA, O'Cleirigh C, Andersen LS, Magidson JF, Lee JS, Bainter SA, Musinguzi N, Simoni J, Kagee A, Joska JA. Treating depression and improving adherence in HIV care with task-shared cognitive behavioural therapy in Khayelitsha, South Africa: a randomized controlled trial. J Int AIDS Soc. 2021 Oct;24(10):e25823. doi: 10.1002/jia2.25823. PMID 34708929
- [Derived] Joska JA, Andersen LS, Smith-Alvarez R, Magidson J, Lee JS, O'Cleirigh C, Safren SA. Nurse-Delivered Cognitive Behavioral Therapy for Adherence and Depression Among People Living With HIV (the Ziphamandla Study): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Feb 3;9(2):e14200. doi: 10.2196/14200. PMID 32012114